CLINICAL TRIAL: NCT03852043
Title: Effect of a HIIT Program Compared to MICT on the Self-esteem, Basal Metabolic Rate and Muscle Mass in Women 18 to 44 Years Old With Overweight or Obesity, Over a Period of 8 Weeks: a Randomized Control Trial.
Brief Title: High-intensity Interval Training on the Self-esteem, Basal Metabolic Rate and Muscle Mass in Overweight Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Associate Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIIT3_AFIS-UdeA
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental)
  Interventions: Behavioral: High-intensity interval training
- Moderate-intensity continuous training (Active Comparator)
  Interventions: Behavioral: Moderate-intensity continuous training

INTERVENTIONS:
Behavioral: High-intensity interval training — The intervals of high intensity are conducted between 90 and 95 % of heart rate maximum (HRmax) and resting between 50 and 60 % of the HRmax 15 loads of 30 seconds at high intensity, with 60 seconds of recovery at loads of moderate intensity.
  Arms: High-intensity interval training
Behavioral: Moderate-intensity continuous training — The continuous training will be carried out at an intensity between 65 and 75% of the HRmax.
  Arms: Moderate-intensity continuous training

SUMMARY:
Overweight and obesity are a public health problem for society, reflected by an increase in its prevalence worldwide, being more frequent in women and related to low levels of self-esteem, accumulation of subcutaneous fat and internal organs, reduction of muscle mass (MM) and basal metabolic rate (BMR). Women are more predisposed to present weight gain because they are metabolically less efficient, have greater food intake, greater physical inactivity, and genetic factors. The different methods of physical training used for weight control are continuous training (CT) and the high-intensity interval training (HIIT). Both CT and HIIT have shown benefits without finding superiority of any of these methods. Nevertheless, there is a trend to the use HIIT programs, since they are more time-efficient and supports their use to induce physiological and metabolic adaptations over time, since this is a barrier to adherence to exercise programs. Overweight and obesity causes individual alterations in body composition and exercise leads to increase in MM, increase in caloric expenditure during the training session and increase in BMR due to the onset of muscle growth, secondary to an increase in the activity of the mitochondrial enzymes (greater mitochondrial biogenesis in the muscle), adaptations that could depend on the type of exercise, its intensity and the volume of it, but it is not clear due to the lack of evidence regarding this.

The primary objective of this study is to demonstrate that a HIIT program of short duration in a real-world setting has a standardized mean difference (SMD) higher than 0.84 in the improvement of self-esteem when comparing with a moderate-intensity continuous training (MICT) in women 18 to 44 years with overweight and obesity and low self-esteem, during eight weeks.

The secondary objective is to demonstrate that a low-volume HIIT in a real-world setting improves MM in 2% compared with MICT during a period of eight weeks in women 18 to 44 years.

DETAILED DESCRIPTION:
Fifty women with low self-esteem will be randomly assigned to one of two training programs (MICT or HIIT) in a real-world setting. Both groups will perform three times a week for eight-weeks on alternate days.

The women in each group will perform three workouts per week for a period of eight weeks. The moderate-intensity continuous training group will perform a training session of 40 min duration at an intensity between 65 and 75% of your HRmax. Women assigned to the group HIIT will perform a training session of 22 minutes of duration by performing intervals of high intensity between 90 and 95 % of the HRmax for 30 seconds in duration and with a recovery of one minute training at moderate intensity is between 50 and 60 % of the HRmax, doing 15 loads of 30 seconds at high intensity, with 60 seconds of recovery between loads at moderate intensity. At the beginning of each training session, both groups will complete strength exercises mainly including large muscle groups (hip, knees, and ankles) with Theraband® (blue color ) for 3 sets of 15 repetitions.

All participants will be evaluated before initiating interventions and upon completion of the training program, after eight weeks, self-esteem will be assessed using the Rosenberg self-esteem scale, determination of anthropometric variables such as weight, height, waist circumference, arterial pressure, body composition by bioimpedance and the basal metabolic rate.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 44 years old, overweighted (BMI ≥ 25 kg / m2) who agree to participate by signing the informed consent, no more than 600 Met / physical activity min / wk (be quantified with the Global Physical Activity Questionnaire - GPAQ), and have less than 30 points on the self-esteem scale.

Exclusion Criteria:

* History of uncontrolled noncommunicable diseases (hypothyroidism, diabetes, asthma and high blood pressure, cardiac arrhythmias), motor disorders or sensitive to hinder the exercise, consumption of anticoagulants, medication altering heart rate (beta-blockers, calcium antagonists, bronchodilators), steroid use, abuse of psychoactive substances, personal history of surgical procedures in the last three months, depressive disorders; pregnancy.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Change in self-esteem | Change from baseline and after 8 weeks
  Self-esteem will be measured by applying the Rosenberg self-esteem scale and according to the scores obtained, the individual will be classified as low self-esteem (<30 points) or normal (> 30 points). The internal consistency of the scale shows a Cronbach's alpha with values ranging between 0.83 and 0.88, and the reliability shows a test-retest correlation of 0.84. Therefore, there is high internal consistency and adequate temporal reliability. Supporting the validity (of construct and known groups) of the instrument.

SECONDARY OUTCOMES:
Change in muscle mass | Change from baseline and after 8 weeks
  Muscle Mass will be quantified through an Omron® HBF510 bioelectrical impedance scale, which has a capacity of 0 to 150 kg, an accuracy of 100 gr for the calculation of weight.

OTHER OUTCOMES:
Change in basal metabolic rate | Change from baseline and after 8 weeks
  Basal metabolic rate will be quantified at the beginning of the study and at the end through a portable gas analyzer model K4b2 (Cosmed Inc, IL, USA), the test will be performed between 7:00 - 7:30 am, the participant must have a fast of at least five hours, and abstaining from consuming products with caffeine and alcoholic beverages 12 hours prior to the evaluation. During the test, the participant must remain seated at rest in an isolated room for 15 minutes. The measurement of the resting metabolic rate will be made during the next 10 minutes in the same position. The criteria to determine a valid measurement will be: the stay in a minimum of 10 minutes in steady state, determined by: discarding the first five minutes of the measurement, reaching a coefficient of variation ≤10% for VO2 and for VCO2 during the ten minutes remaining and a respiratory quotient between 0.7 to 1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Elkin F Arango, MD. MsC, Study Director — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No